CLINICAL TRIAL: NCT07347327
Title: The Effect of Dual-target tACS Combined With Speech Training on Repetition Disorder After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ke Dong, MD (Other)
Responsible Party: Sponsor-Investigator, Ke Dong, MD, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Nos.82102648
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real group (Experimental): dual-target tACS on auditory and motor brain area at a frequency of 8 Hz,with individualized current intensity, delivered for 20 minutes.
  Interventions: Behavioral: speech training; Other: real tACS
- sham group (Sham Comparator): sham tACS except for turning down the current intensity to zero during the 20-minute period, all other parameters are identical to those in real group.
  Interventions: Behavioral: speech training; Other: sham tACS

INTERVENTIONS:
Behavioral: speech training — speech training(especially repetition training) synchronized with tACS stimulation
Other: real tACS — dual-target tACS on auditory and motor brain area at a frequency of 8 Hz,with individualized current intensity, delivered for 20 minutes.
  Arms: real group
Other: sham tACS — except for turning down the current intensity to zero during the 20-minute period, all other parameters are identical to those in real group.
  Arms: sham group

SUMMARY:
This clinical trial aims to study whether dual-target transcranial alternating current stimulation (tACS) applied to the auditory and motor brain region can improve repetition disorder in people with stroke, and to evaluate the safety of tACS. The main goals are to answer the following questions:

1. Can dual-tACS stimulation of the auditory and motor brain area improve repetition functions in people with aphasia after stroke?
2. Can it improve the integration of auditory information and speech motor control during communication?

Researchers will compare the effects of real tACS versus sham (placebo) stimulation to see if real stimulation leads to better outcomes in aphasia patients.

Participants will:

1. Receive one extra 20-minute session of either real or sham tACS each day for 10 days
2. Attend clinic visits before and after 10-days stimulation for clinical assessments(WAB) and fNIRS recording related brain activity

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria for hemorrhagic or ischemic stroke in the Chinese Guidelines for the Prevention and Treatment of Cerebrovascular Diseases(2nd edition), with the first onset, single hemisphere stroke, and confirmed by CT or MRI,course of diease 1-6 months;
* Age ranging from 30 to 80 years old;
* Native language is Mandarin or Cantonese;
* Right-handed;
* Diagnosed with aphasia by the Western Aphasia Battery (WAB) scale;
* Able to cooperate in completing the speech repetition test;
* Normal hearing.

Exclusion Criteria:

* Currently receiving non-invasive brain stimulation treatment;
* Lesions involving the Broca or STG brain regions;
* History of epilepsy, mental illness,or other neurological or mental disorders;
* Any contraindications for transcranial electrical stimulation.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-26 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Western Aphasia Battery (WAB) score | Baseline and 10-days
  Western Aphasia Battery (WAB) score：0-100，higher score means better language function

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Medicine, The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China